CLINICAL TRIAL: NCT06676475
Title: Comparison of the Effectiveness of Botulinum Toxin and Magnesium Sulfate Injections in the Treatment of Myofascial Trigger Points in the Masseter Muscle Randomized Controlled Clinical Trial
Brief Title: Comparison Between Botox and Magnesium Sulfate Effect in Treatment of Myofascial Pain Trigger Points Within the Masseter Muscle
Acronym: MPS MTrPs BTA
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Mayada tarek, B.D.S. Faculty of Oral and Dental Surgery, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200036178
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Myofacial Pain; Trigger Points, Myofascial
Keywords: myofascial pain; masseter trigger point; MPS; MTrPs; MgSO4 in myofascial trigger points; BTA in myofascial trigger points; Botox in masseter trigger points; magnesium sulfate in masseter trigger points
MeSH Terms: conditions — Facial Pain | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I: Patients will receive Magnesium Sulfate injection into trigger points (Experimental)
  Interventions: Drug: MgSO4
- Group II: Patients will receive Botulinum Toxin into trigger points (Active Comparator)
  Interventions: Drug: BOTOX-A
- Group III: Patients will receive Saline injection into trigger points (Placebo Comparator)
  Interventions: Drug: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Drug: MgSO4 — 2ml MgSo4 (Magnesium sulfate sterile ampoule 10 ml, 100 mg/ml = 0.41 mMol/ml. Egyptian Int. Pharmaceutical Industries Co., Egypt).
  Arms: Group I: Patients will receive Magnesium Sulfate injection into trigger points
Drug: BOTOX-A — 2ml of BTX
  Arms: Group II: Patients will receive Botulinum Toxin into trigger points
Drug: Saline (NaCl 0,9 %) (placebo) — 2 ml of saline
  Arms: Group III: Patients will receive Saline injection into trigger points

SUMMARY:
The goal of this randomized clinical trial is to compare the effectiveness of Botulinum toxin type A, magnesium sulfate and saline injections in treatment of the masseter muscle trigger points, in patients between 16 - 50 years old with myofascial pain with masseter muscle trigger points. The main questions it aims to answer are:

* which treatment has longer effect of pain release with the least possible side effects and recurrence rate?
* Which treatment has greater impact on improving patient's quality of life? Researchers will compare Botulinum toxin type A, magnesium sulfate to a placebo saline injections in treatment of the masseter muscle trigger points Participants will attend to the clinic 4 times
* 1st visit will include taking preoperative records and treatment injection
* 2nd visit will be follow up and taking records after 1 month
* 3rd visit will be follow up and taking records after 3 months
* 4th visit will be follow up and taking records after 6 months

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is common syndrome in patients with musculoskeletal pain problems. It's a pain condition originating from muscle and surrounding fascia. Patient usually complains from localized pain in a certain area or referred pain of various patterns. On physical examinations, trigger points (TrPs) may reveal on the involved muscles. (Tantanatip, Chang,2018). TrPs are usually palpable and hyperirritable nodule found within a taut band of muscle. By Stimulating these points, two characteristic phenomena are produced: sudden contractions of the taut band and referred pain, which is known as the local twitch response (LTR). Active MTrPs usually produce pain spontaneously, and sometimes referred pain, while Latent MTrPs produce referred pain in response to the applied pressure, but not spontaneously (Simons, D.G, 2004).

Multiple factors can contribute to MPS. The risk factors are; Traumatic events, ergonomic factors (e.g., overuse activities, abnormal posture, Structural factors (e.g., spondylosis, scoliosis, osteoarthritis), systemic factors (e.g., hypothyroidism, vitamin D deficiency, iron deficiency). (Saxena,et al,2015), however Intramuscular injections are considered the first-line treatment for myofascial TrPs(Yilmaz, et al 2021). Injections could be wet as local anesthetic agents, steroid, platelet rich plasma, saline or botulinum toxin, or it could be dry by dry needling without solutions MPS is a result of inappropriate activity of acetylcholine (ACh) at the neuromuscular junction, producing a sustained contraction of the sarcomere. The ACh-related effects are relevant to the taut band development, which leads to increasing the local energy demand or energy crisis (Simons, D.G, 2004). The pain in the local muscle occurs secondary to the substances released from the damaged muscle, and from the extracellular fluid around the TrP, such as protons (H+) on acid-sensing ion channels which occurs in ischemia and in exercise. In these metabolic conditions, sensitizing amines may be released stimulating the nociceptors and giving rise to pain. Therefore, MTrPs are better defined by two phenomena: altered ACh activity and nociceptive stimulation (Sluka, Kalra, Moore,2001). The fact of myofascial muscles are a part of the stomatognathic system, any imbalance in this system could have a disturbing impact on its function such as mastication, posture and non-physiological occlusion, affecting the patient's quality of life (Fiorillo, 2020).

Botulinum toxin type A is a neurotoxin used to reduce excessive muscle contraction. Its produced by gram-positive, anaerobic, spore-forming bacilli known as Clostridium botulinum which is widely distributed in aquatic and soil environments. (Tiwari,Nagalli 2024). Botulinum toxin inhibits neurotransmission at the neuromuscular junction. Several transport proteins participate in the process by which ACh is released; these proteins aggregate to form the SNARE complex (Soluble NSF (N-Ethylmaleimide-Sensitive Factor) Attachment Protein Receptor, responsible for fusion of the vesicles of ACh with the membrane and the subsequent release of the neurotransmitter. The heavy chain of the toxin has a high affinity for the membrane receptors and, once bound, BTA undergoes endocytosis. The light chain is released within the cell, where it acts as a zinc-dependent endoprotease. After cleavage of one of the proteins of the SNARE complex by BTA, the complex does not form and ACh is not released. (Aikawa,et al , 2006) Magnesium sulfate (MgSO4) is commonly used as analgesics for treatment of musculoskeletal problems, snice having muscle relaxant and vasodilator properties. (Ibrahim, Raoof, Mosaad,2021). These properties can likely be attributed to its ability to block presynaptic acetylcholine discharge from neuromuscular and sympathetic junctions (Dahle, et al ,1995). Therefore, MgSo4 injections are an effective treatment modality for myofascial TrPs of the masseter muscle. It helps in reducing the pain and improving the maximum mouth opening, in addition to the quality of patient's life. (Refahee, Mahrous, Shabaan,2022)

Intervention After the MTP is located and the overlying skin had been disinfected with alcohol, the taut muscle band is pinched between the thumb and index finger, and the needle is inserted 1-2 cm away from the targeted MTP at an angle of 30º to the skin. A negative aspiration should be performed to prevent any intravascular injections (Taşkesen, Cezairli, 2023). Group 1: 2ml MgSo4 (Magnesium sulfate sterile ampoule 10 ml, 100 mg/ml = 0.41 mMol/ml. Egyptian Int. Pharmaceutical Industries Co., Egypt). Group 2: 2ml of BTX and Group 3: 2 ml of saline

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with orofacial pain and trigger points in the masseter muscle unilaterally or bilaterally for at least period 6 months other criteria
* Definite diagnosis of myofascial pain based on the DC/TMD criteria with a referral
* Presence of one or more unilateral or bilateral trigger points in the masseter muscle
* No history of any invasive procedures of the related masseter muscle (Taşkesen, Cezairli, 2023.)

Exclusion Criteria:

* Any painful conditions (other than myofascial trigger points) affecting the orofacial region
* Any systemic diseases that could affect masticatory function (e.g., rheumatoid arthritis and epilepsy
* Pregnancy and lactation. (Refahee, Mahrous, Shabaan,2022)

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluating pain | preoperative - post operative - 1 , 3 ,6 months follow up
  Pain will be recorded with a visual analog scale (VAS of 0-10, with zero being no pain and 10 the worst pain possible)

SECONDARY OUTCOMES:
Pain-free maximum mouth opening (MMO) | preoperative - post operative - 1 , 3 ,6 months follow up
  Pain-free MMO will be measured as the distance between the incisal edges of the upper and lower incisors. Three measurements will be performed, and their average was recorded (Taşkesen, Cezairli, 2023).
Muscle health and activity measured using electromyography | preoperative - post operative - 1 , 3 ,6 months follow up
  Muscle health and activity measured using electromyography, EMG can provide valuable insights into altered muscle activity patterns and help in the diagnosis and management of MPDS through readings (Zieliński, et al, 2021).
The quality of life will be assessed using the Oral Health Impact Profile questionnaire (OHIP-14) | preoperative - post operative - 1 , 3 ,6 months follow up
  The quality of life will be assessed using the Oral Health Impact Profile questionnaire (OHIP-14) containing 14 questions divided into seven domains of oral health. The participant will be asked to score each question using a scale from 1 to 5 [never (score 0); hardly ever (score 1); occasionally (score 2); fairly often (score 3); and very often (score 4)], and the sum of all 14 items was calculated. The OHIP score could range from 0 to 56 units, with the former indicating no problems and higher scores representing greater impairment of quality of life (Slade and Spencer, 1994).

CONTACTS AND LOCATIONS:
Locations (1):
- Misr university for science and technology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zielinski G, Bys A, Szkutnik J, Majcher P, Ginszt M. Electromyographic Patterns of Masticatory Muscles in Relation to Active Myofascial Trigger Points of the Upper Trapezius and Temporomandibular Disorders. Diagnostics (Basel). 2021 Mar 24;11(4):580. doi: 10.3390/diagnostics11040580. PMID 33805008
- [Background] Yilmaz O, Sivrikaya EC, Taskesen F, Pirpir C, Ciftci S. Comparison of the Efficacy of Botulinum Toxin, Local Anesthesia, and Platelet-Rich Plasma Injections in Patients With Myofascial Trigger Points in the Masseter Muscle. J Oral Maxillofac Surg. 2021 Jan;79(1):88.e1-88.e9. doi: 10.1016/j.joms.2020.09.013. Epub 2020 Sep 14. PMID 33045182
- [Background] Taskesen F, Cezairli B. The effectiveness of the masseteric nerve block compared with trigger point injections and dry needling in myofascial pain. Cranio. 2023 Mar;41(2):96-101. doi: 10.1080/08869634.2020.1820686. Epub 2020 Sep 16. PMID 32935643
- [Background] Tantanatip, A. and Chang, K.V., 2018. Myofascial pain syndrome.
- [Background] Sluka KA, Kalra A, Moore SA. Unilateral intramuscular injections of acidic saline produce a bilateral, long-lasting hyperalgesia. Muscle Nerve. 2001 Jan;24(1):37-46. doi: 10.1002/1097-4598(200101)24:13.0.co;2-8. PMID 11150964
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Simons DG. Review of enigmatic MTrPs as a common cause of enigmatic musculoskeletal pain and dysfunction. J Electromyogr Kinesiol. 2004 Feb;14(1):95-107. doi: 10.1016/j.jelekin.2003.09.018. PMID 14759755
- [Background] Saxena A, Chansoria M, Tomar G, Kumar A. Myofascial pain syndrome: an overview. J Pain Palliat Care Pharmacother. 2015 Mar;29(1):16-21. doi: 10.3109/15360288.2014.997853. Epub 2015 Jan 5. PMID 25558924
- [Background] Refahee SM, Mahrous AI, Shabaan AA. Clinical efficacy of magnesium sulfate injection in the treatment of masseter muscle trigger points: a randomized clinical study. BMC Oral Health. 2022 Sep 19;22(1):408. doi: 10.1186/s12903-022-02452-3. PMID 36123724
- [Background] Pihut M, Ferendiuk E, Szewczyk M, Kasprzyk K, Wieckiewicz M. The efficiency of botulinum toxin type A for the treatment of masseter muscle pain in patients with temporomandibular joint dysfunction and tension-type headache. J Headache Pain. 2016;17:29. doi: 10.1186/s10194-016-0621-1. Epub 2016 Mar 24. PMID 27011213
- [Background] Nitecka-Buchta A, Walczynska-Dragon K, Batko-Kapustecka J, Wieckiewicz M. Comparison between Collagen and Lidocaine Intramuscular Injections in Terms of Their Efficiency in Decreasing Myofascial Pain within Masseter Muscles: A Randomized, Single-Blind Controlled Trial. Pain Res Manag. 2018 Jun 3;2018:8261090. doi: 10.1155/2018/8261090. eCollection 2018. PMID 29973970
- [Background] Ibrahim NA, Abdel Raoof NA, Mosaad DM, Abu El Kasem ST. Effect of magnesium sulfate iontophoresis on myofascial trigger points in the upper fibres of the trapezius. J Taibah Univ Med Sci. 2021 Jan 19;16(3):369-378. doi: 10.1016/j.jtumed.2020.12.015. eCollection 2021 Jun. PMID 34140864
- [Background] Fiorillo L. Spine and TMJ: A Pathophysiology Report. J Funct Morphol Kinesiol. 2020 Mar 30;5(2):24. doi: 10.3390/jfmk5020024. PMID 33467240
- [Background] Dahle LO, Berg G, Hammar M, Hurtig M, Larsson L. The effect of oral magnesium substitution on pregnancy-induced leg cramps. Am J Obstet Gynecol. 1995 Jul;173(1):175-80. doi: 10.1016/0002-9378(95)90186-8. PMID 7631676
- [Background] Blanco-Rueda JA, Lopez-Valverde A, Marquez-Vera A, Mendez-Sanchez R, Lopez-Garcia E, Lopez-Valverde N. Preliminary Findings of the Efficacy of Botulinum Toxin in Temporomandibular Disorders: Uncontrolled Pilot Study. Life (Basel). 2023 Jan 28;13(2):345. doi: 10.3390/life13020345. PMID 36836702
- [Background] Aikawa Y, Lynch KL, Boswell KL, Martin TF. A second SNARE role for exocytic SNAP25 in endosome fusion. Mol Biol Cell. 2006 May;17(5):2113-24. doi: 10.1091/mbc.e06-01-0074. Epub 2006 Feb 15. PMID 16481393